CLINICAL TRIAL: NCT01725334
Title: Deep Brain Stimulation for the Management of Treatment Refractory Negative Symptoms in Schizophrenia
Brief Title: Deep Brain Stimulation (DBS) for the Management of Treatment Refractory Negative Symptoms in Schizophrenia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other); Schizophrenia Society of Ontario (Other)
Responsible Party: Principal Investigator, Z. J. Daskalakis, Chair, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 078/2011
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Schizophrenia; Negative Type
Keywords: Schizophrenia; Negative Symptoms; Treatment Resistance; Deep Brain Stimulation; Electrical Stimulation; Mental Disorders; Brain Diseases; Neurologic Manifestations; Signs and Symptoms
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Brain Diseases; Neurologic Manifestations; Signs and Symptoms | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nucleus Accumbens/Ventral Striatum (NAcc/VS) Stimulation (Experimental): The first 3 patients will have the DBS device target the NAcc/VS, which has been found to be hypoactive in patients with primarily negative symptoms.
  Interventions: Procedure: Deep Brain Stimulation
- Ventral Tegmental Area (VTA) Stimulation (Experimental): For 3 patients, the DBS device will target the VTA, which has been found to be hypoactive in patients with primarily negative symptoms.
  Interventions: Procedure: Deep Brain Stimulation

INTERVENTIONS:
Procedure: Deep Brain Stimulation — Deep Brain Stimulation (DBS) is a surgical procedure involving the implantation of a thin flexible wire called a lead. This device sends mild electric signals to an area of the brain. This study targets two different areas that we believe may be responsible for negative symptoms observed in patients with schizophrenia. There are two stages to DBS: (1) Insertion of the DBS electrodes (2) The connection of these electrodes to a battery under the collarbone.
  Other Names: DBS

SUMMARY:
Schizophrenia is a complex, challenging, and heterogeneous psychiatric condition, affecting up to 0.5% of the population and responsible for nearly 2% of all Canadian health-care expenditure. Much of the morbidity of the illness is related to its negative symptoms, including amotivation, asociality, anhedonia and flattened emotional affect, which lead to functional impairment and withdrawal from social and occupational domains. In contrast to positive symptoms, such as hallucinations and delusions, there are currently no effective treatments for negative symptoms, which experts recognize are largely responsible for the long-term disability of a majority of patients with schizophrenia. Advances in neuroscience have allowed a greater understanding of negative symptoms and have identified key structures and circuits believed to generate and maintain them. Here, we propose the application of a targeted therapy, deep brain stimulation, to alter the circuits driving negative symptoms.

DETAILED DESCRIPTION:
Schizophrenia is a public health challenge with a large proportion of patients suffering from predominantly negative symptoms and who derive no benefit from currently available treatments. Advances in neuroscience have allowed a greater understanding of negative symptoms and have identified key structures and circuits believed to generate and maintain them. Here, we propose the application of a targeted therapy, deep brain stimulation (DBS), to alter the circuits driving negative symptoms. This is a phase I, non-blinded, non-randomized, pilot trial, exploring the safety and efficacy of DBS in patients with refractory negative symptoms of schizophrenia. Patients must be identified and approached by their treating psychiatrist regarding this study. Patients will be given several opportunities to review the study details with the investigators before the informed consent is presented. All eligible patients will also be reviewed by an independent non-study affiliated psychiatrist for confirmation of their diagnosis and assessment of study eligibility. The total study duration will be one year for each patient, who will undergo regular imaging and psychiatric analyses.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients between the age of 25-65
* DSM IV-TR diagnosis of Schizophrenia Predominant Negative Subtype, as determined by the SANS and the Schedule for the Deficit Syndrome (SDS)
* Greater negative than positive scores on the Positive and Negative Symptoms of Schizophrenia Scale (PANSS)
* Confirmation of diagnosis by independent, non-study affiliated psychiatrist
* Disease duration of > 5 years
* Failure of medical therapy, defined as follows:
* Failure of a minimum of three anti-psychotic treatments for specifically negative symptoms of schizophrenia (including clozapine)
* No underlying neurological disease - No other active Axis I or Axis II co-morbidity that is the focus of clinical attention
* Able to give informed consent: i)Deemed competent by two independent psychiatrists (one study psychiatrist and one non-study psychiatrist); ii) Score of > 70 on MacCat-CR
* Able to comply with all testing and follow-up visit requirements defined by the Study Protocol
* Mini mental status examination (MMSE)score > 25
* Pre-menopausal women must agree to use acceptable methods of birth control (radiation risk of PET)

Exclusion Criteria:

* Alcohol or substance dependence or abuse within 6 months, excluding nicotine or caffeine.
* Current suicidal ideation, plan or intent for self-harm.
* A suicide attempt in the past 1 year
* Diagnosis of Major Depressive Disorder or Bipolar Depression
* Major medical illness, cardiac pacemaker/defibrillator, and other implanted stimulator
* Likely to relocate or move to a location distant from the study site within one year of enrollment
* Any contraindication to MRI or PET scanning
* Inability to provide consent, as well as an inability to appreciate the details and risk of the trial's procedures; competence will be assessed by two independent psychiatrists (one study psychiatrist, and one non-study psychiatrist)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Schedule for the Assessment of Negative Symptoms (SANS) | Change from baseline (pre-operative) SANS scores at one-year follow-up
  Assessment of primary and enduring negative symptoms consisting of affective blunting, alogia, avolition, anhedonia/asociality and impairments in attention.
  It is numerically graded on a scale from 0 to 5; 0 being not at all present and 5 being severe.

CONTACTS AND LOCATIONS:
Overall Officials: Zafiris J Daskalakis, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.ca/en/research/Pages/research.aspx